CLINICAL TRIAL: NCT05320744
Title: Evaluation the Effect of Angle of Impaction, Impaction Depth, and Bone Density on Surgical Difficulty of Impacted Mandibular Third Molar by Using Orthopantomography
Brief Title: the Relationship Between Various Clinical Variables and Surgical Difficulty of Patients Have Impacted Lower Third Molar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed, Principal Investigator, University of Baghdad
Other Study IDs: impacted lower third molar
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgical extraction of impacted lower third molar — surgical removal of impacted third molar under local anesthesia.

SUMMARY:
This study is to evaluate the effect of angle of impaction, impaction depth, and bone density on surgical difficulty of impacted lower third molar, by measuring the angle of impaction, the depth of impaction (Winter's Red line), and bone density (gonial, and antegonial indices) preoperatively by using panoramic radiograph and to correlate the angle, the depth of impaction, and bone density with the surgical difficulty by operation time and surgical technique.

DETAILED DESCRIPTION:
* All patients will provide detailed medical history and will sign a written informed consent. Oral hygiene instruction, scaling, and root planing.
* Panoramic radiograph will be taken for every patient, It will be used for measuring the angle of impaction along the lamina dura of the lower second and third molar and measuring impaction depth (Winter's Red line) by using software (planmeca romexis). The same software will be used to measure gonial index and antegonial angle as indices of bone density.
* All patients will have mouth rinsing with 0.2% chlorhexidine digluconate for 1 minute.

Surgical Procedure

* After administration of local anesthesia, full thickness enveloped or triangular flap incision according to the surgical principles.
* Flap reflection with periosteal elevator and retraction.
* Bone removal (if required) by using a slow speed, high torque surgical handpiece with sharp bur with copious normal saline irrigation.
* Tooth sectioning (if required) by using sharp diamond bur with saline irrigation.
* Tooth extraction by using appropriate elevator. .The operative difficulty will be determined by the surgical techniques of the extraction and the duration of extraction. With respect to the surgical technique the degree of difficulty is considered low when the extraction is performed by elevator alone, moderate when bone removal (ostectomy) is required, and high when ostectomy and tooth sectioning is required for tooth extraction.

For the duration of surgery, the difficulty is considered low when the duration of surgical extraction is less than 15 minutes, moderate when the duration is 15-30 minutes, and high when the duration is more than 30 minutes.

* Irrigation and cleaning of surgical site and removing remaining follicle if present.
* Bone smoothing with bone file and irrigation with saline.
* Flap Suturing with black silk suture 3/0.
* Ask the patient to bite on wet gauze.
* Instruction and medication (analgesic and antibiotic if required).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients over 18 years old of either gender.
2. Patients who have mesioangular or horizontal impacted mandibular third molar.
3. Presence of mandibular second molar.
4. Ability to tolerate surgical procedure.

Exclusion Criteria:1. Patients with vertically and distoangularlly impacted teeth.

2. Patients with uncontrolled systemic diseases. 3. Patients with history of chemotherapy or radiotherapy therapy to the head and neck region.

4. Acute infection at the surgical site at time of operation. 5. The presence of cysts or tumors associated with the impacted teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include a minimum of 50 patients indicated for surgical removal of impacted mandibular third molars at Baghdad college of dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Angle of impaction | preoperative
  is measured along the lamina dura of lower second and third molar by using Planmeca Romexis Software.
Winter Red line | preoperative
  is measured by drawing perpendicular line from amber line to the point of application of dental elevator by using Planmeca Romexis Software
Gonial index | preoperative
  is measurement of mandibular cortical thickness by using bisectrix the gonial angle by using Planmeca Romexis Software
Antegonial angle | preoperative
  is the measurement of the mandibular cortical thickness measured on the line perpendicular to the mandibular cortex at the intersection with the tangent line to the anterior border of the ramus by using Planmeca Romexis Software
operative difficulty | intraoperative
  determined by the surgical techniques of the extraction and the duration of extraction according to Pernambuco difficulty scale

CONTACTS AND LOCATIONS:
Overall Officials: Salwan Y. Bede, F.I.B.M.S, Study Chair — Baghdad college of dentistry/ Department of oral and maxillofacial surgery
Locations (1):
- university of Baghdad/ Baghdad college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
all the results
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] de Carvalho RWF, Vasconcelos BC. Pernambuco index: predictability of the complexity of surgery for impacted lower third molars. Int J Oral Maxillofac Surg. 2018 Feb;47(2):234-240. doi: 10.1016/j.ijom.2017.07.013. Epub 2017 Aug 14. PMID 28818641
- [Result] Zhang X, Wang L, Gao Z, Li J, Shan Z. Development of a New Index to Assess the Difficulty Level of Surgical Removal of Impacted Mandibular Third Molars in an Asian Population. J Oral Maxillofac Surg. 2019 Jul;77(7):1358.e1-1358.e8. doi: 10.1016/j.joms.2019.03.005. Epub 2019 Mar 14. PMID 30959010